CLINICAL TRIAL: NCT00638963
Title: Temozolomide in Metastatic Breast Cancer Patients at High Risk of Brain Recurrence: Impact on the Incidence of Brain Metastases (STOP)
Brief Title: Temozolomide as a Prophylaxis Against Brain Recurrence in Participants With Metastatic Breast Cancer (P05225 AM2)
Acronym: STOP
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to poor accrual
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P05225; 2007-005491-14 (EudraCT Number)
Record Dates: First submitted 2008-01-10; First posted 2008-03-19 (Estimated); Results first posted 2011-07-22 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Breast Neoplasm; Brain Neoplasm; Second Neoplasm
MeSH Terms: conditions — Breast Neoplasms; Brain Neoplasms; Neoplasms, Second Primary | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Temozolomide (Experimental)
  Interventions: Drug: temozolomide
- Observational (No Intervention)

INTERVENTIONS:
Drug: temozolomide — Capsules to equal 75 mg/m^2, orally, daily for 6 weeks, in 3 eight-week cycles
  Arms: Temozolomide

SUMMARY:
The purpose of this study is to determine whether temozolomide can be used as a prophylaxis against brain recurrence in participants with metastatic breast cancer.

DETAILED DESCRIPTION:
Breast cancer is the second most common cause of brain metastases. Overall survival after the development of brain metastases tends to be poor (6-8 months). Over-expression of Human Epidermal Growth Factor Receptor 2 (HER-2/neu), negative estrogen receptor, and young age at diagnosis seem to be indicators of high risk for brain metastases. Temozolomide may be a good candidate for prophylactic chemotherapy because of its ability to cross the blood-brain-barrier, achieving high concentrations in the central nervous system (CNS).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of metastatic breast cancer.
* Participants must have completed first line of metastatic chemotherapy and have achieved complete or partial response or disease stability for at least 6 months from the first confirmation of disease stabilization.
* No clinical sign of brain progression.
* At least one of the following 3 conditions: HER2 +++, Young age (< 50 years), and/or estrogen receptor (ER)-/progesterone receptor (PgR)-
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
* Life expectancy ≥3 months.
* Neutrophils ≥1.5 x 10^9/L, platelets ≥100 x 10^9/L, hemoglobin ≥9 g/dL, lymphocytes ≥1 x 10^9/L.
* Bilirubin level either normal or <1.5 x ULN (upper limit of normal).
* AST (aspartate aminotransferase) and ALT (alanine aminotransferase) ≤2.5 x ULN (≤5 x ULN if liver metastases are present).
* Serum creatine <1.5 x ULN.
* Effective contraception if the risk of conception exists.

Exclusion Criteria:

* Concurrent chronic systemic immune therapy not indicated in the study protocol.
* Any investigational agent(s) within 4 weeks prior to entry.
* Participants that have completed 2nd, 3rd, or 4th line metastatic chemotherapy or participant in active chemotherapy treatment.
* Clinically relevant coronary artery disease or a history of a myocardial infarction within the last 12 months.
* Acute or sub acute intestinal occlusion or history of inflammatory bowel disease.
* Known Grade 3 or Grade 4 allergic reaction to any of the components of the treatment.
* Known drug abuse/alcohol abuse.
* Legal incapacity or limited legal capacity.
* Medical or psychological condition which in the opinion of the investigator would not permit the participant to complete the study or sign meaningful informed consent.
* Women who are pregnant or breastfeeding.
* Any concurrent malignancy other than non-melanoma skin cancer, or carcinoma in situ of the cervix (participants with a previous malignancy but without evidence of disease for ≥5 years will be allowed to enter the trial).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-10-02 (Actual); Primary Completion 2010-06-30 (Actual); Study Completion 2010-06-30 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Groups:
- Observational: No temozolomide treatment
Period: Overall Study
Arm/Group | Temozolomide | Observational
Started | 3 (Received randomized treatment assignment) | 3 (Received randomized treatment assignment)
Completed | 2 (including follow-up at Week 38 & Week 52) | 3 (including follow-up at Week 38 & Week 52)
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Temozolomide | Observational | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Italy | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With Recurrence of Brain Metastases
Description: The analysis could not be performed due to low enrollment.
Time Frame: 1 Year
Arm/Group | Temozolomide | Observational
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number of Days With Progression-free Survival (PFS)
Description: PFS was defined as the time interval from randomization to objective tumor progression or death from any cause.
  The analysis could not be performed due to low enrollment.
Time Frame: 24, 38, and 52 weeks
Arm/Group | Temozolomide | Observational
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Days With Disease-free Survival (DFS)
Description: DFS was defined as the time interval from randomization to any relapse (loco-regional, contra-lateral, and/or distant).
  The analysis could not be performed due to low enrollment.
Time Frame: 24, 38, and 52 weeks
Arm/Group | Temozolomide | Observational
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Days With Distant Disease-free Survival (DDFS)
Description: DDFS was defined as the time interval from randomization to only distant metastases (for example, bone, visceral organ, brain).
  The analysis could not be performed due to low enrollment.
Time Frame: 24, 38, and 52 weeks
Arm/Group | Temozolomide | Observational
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Days With Brain Recurrence-free Survival (BRFS)
Description: BRFS was defined as the time interval from randomization to the appearance of brain metastases.
  The analysis could not be performed due to low enrollment.
Time Frame: 24,38, and 52 weeks
Arm/Group | Temozolomide | Observational
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Number of Days on Temozolomide Treatment
Description: This outcome measure was only applicable to the temozolomide arm; the observation arm was therefore not analyzed.
Time Frame: Baseline to 24 Weeks
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Temozolomide
Number analyzed (Participants) | 3
Days | 75 (65.82) [1 to 127]

7. Secondary Outcome: Total Dose of Temozolomide Taken
Description: This outcome measure was only applicable to the temozolomide arm; the observation arm was therefore not analyzed.
Time Frame: Baseline to 24 Weeks
Measure: Mean (Standard Deviation); unit: Milligrams
Arm/Group | Temozolomide
Number analyzed (Participants) | 3
Milligrams | 9791.9 (8732.0)

8. Secondary Outcome: Number of Participants Who Had at Least One Dose Reduction During Treatment
Description: This outcome measure was only applicable to the temozolomide arm; the observation arm was therefore not analyzed.
Time Frame: Baseline to 24 Weeks
Measure: Number; unit: Participants
Arm/Group | Temozolomide
Number analyzed (Participants) | 3
Participants | 3

9. Secondary Outcome: Number of Participants Who Had at Least One Treatment Omission During Treatment
Description: This outcome measure was only applicable to the temozolomide arm; the observation arm was therefore not analyzed.
Time Frame: Baseline to 24 Weeks
Measure: Number; unit: Participants
Arm/Group | Temozolomide
Number analyzed (Participants) | 3
Participants | 2

10. Secondary Outcome: Number of Participants Who Completed the Third Cycle of Treatment
Description: This outcome measure was only applicable to the temozolomide arm; the observation arm was therefore not analyzed.
Time Frame: Baseline to 24 Weeks
Measure: Number; unit: Participants
Arm/Group | Temozolomide
Number analyzed (Participants) | 3
Participants | 2

ADVERSE EVENTS:
Arm/Group | Temozolomide | Observational
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 2/3 | 2/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temozolomide (N=3) | Observational (N=3)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (6) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (3) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The primary outcome measure and the survival analyses could not be analyzed due to the low enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The principal investigator (PI) agrees not to publish or publicly present any interim results of the Study without prior written consent of the sponsor. The PI further agrees to provide 45 days written notice to the sponsor prior to submission for publication or presentation to permit the sponsor to review copies of abstracts or manuscripts for publication in accordance with provisions of laws related to protection of sensitive personal data and patentability of inventions.